CLINICAL TRIAL: NCT04932954
Title: Immunohematology in COVID-19 Patients: A Hospital-based Retrospective Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: LI YAN (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Henan University of Science and Technology (Other)
Responsible Party: Sponsor-Investigator, LI YAN, professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ-IRB20210603
Record Dates: First submitted 2021-06-17; First posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Covid19
Keywords: Immunohematology; Blood group; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a hospital-based retrospective cohort study and the Immunohematologic characteristics of COVID-19 patients will be investigated systematically.

DETAILED DESCRIPTION:
This is a hospital-based retrospective cohort study and the Immunohematologic characteristics of COVID-19 patients will be investigated systematically. In this study, we will seek to understand the association between SARS-CoV-2 infection and blood groups and explore the Anti-A and Anti-B effects in COVID-19 patients with graded severity. We will analyze the transfusion requirement and the clinical recurrences of COVID-19 patients. The discrepancy of blood group phenotypes in COVID-19 patients with graded severity will be also analyzed on the molecular level. This retrospective cohort study was conducted using electronic health recording data in Tongji Hospital. The clinical characteristics for all eligible patients will be retrieved. The records will be verified to avoid possible bias. Data collection was carried out independently by two investigators and reviewed by two different investigators.

ELIGIBILITY:
Inclusion Criteria:

* The patients who were diagnosed with COVID-19 following the WHO interim guidelines (https://www.who.int/publications-detail/clinical-management-of-severe-acute-respiratory-infection-when-novelcoronavirus-(ncov)-infection-is-suspected. 2020.)

Exclusion Criteria:

* Male or female patients <18 years of age

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients were diagnosed with COVID-19 following the WHO interim guidelines and admitted for treatment in Tongji hospital. The admission dates were January 01 2020 to April 01, 2021. Male or female patients <18 years of age were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
ABO and Rh distribution | 1 year
  ABO and Rh phenotype distribution refers to the phenotype frequency of the ABO and Rh subtypes in severe and non-severe COVID-19 patients
ABO antibody titers | 1 year
  ABO antibody titers refers to both anti-A and anti-B antibodies in severe and non-severe COVID-19 patients

SECONDARY OUTCOMES:
Transfusion incidence | 1 year
  Transfusion incidence refers to the number of COVID-19 hospitalized patients who received transfusion
Patients with coagulopathy | 1 year
  Patients with coagulopathy refers to patients hospitalized with Covid-19 to develop coagulopathy
Leukocyte and neutrophil counts | 1 year
  Leukocyte and neutrophil counts refer to the number of Leukocyte and neutrophil COVID-19 hospitalized patients with graded severity
outcomes of SARS-CoV-2 infection | 1 year
  outcomes of SARS-CoV-2 infection refer to the intubation and death in SARS-CoV-2 infected patients
Polymorphism of ABO blood group | 1 year
  Polymorphism of ABO blood group refers to the variations and alleles of the ABO gene in COVID-19 patients

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China